CLINICAL TRIAL: NCT01829633
Title: Anatomic and Clinical Long-term Follow-up of Conservatively Treated Rotator Cuff Tears
Status: Completed | Type: Observational
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Principal Investigator, Stefan Moosmayer, MD, PhD, Vestre Viken Hospital Trust
Other Study IDs: 29144/3/LT; 2011/1931 (Other: Regional Committees for Medical and Health Research Ethics)
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Full-thickness Rotator Cuff Tears
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Rotator cuff tears: Patients who were diagnosed with a symptomatic full-thickness tear of the rotator cuff. Tear examination by sonography and MRI showed a repairable tear. All patients were initially treated conservatively by physiotherapy.
  Interventions: Procedure: Physiotherapy

INTERVENTIONS:
Procedure: Physiotherapy — Shoulder physiotherapy with exercises

SUMMARY:
Study population: Patients who have been treated with physiotherapy for a potentially repairable rotator cuff tear in the period from 2002 to 2005.

Study Method: At the time of diagnosis (2002 to 2005) all study patients were examined clinically, sonographically and by MRI. Some patients also completed a shoulder score. All study patients will now be reexamined, 8 to 10 years after they were diagnosed. Reexamination includes history taking, clinical examination, completion of three shoulder scores (two shoulder specific scores, one general health score), Sonography and MRI. Findings of interest are

* the number of relapses during follow-up,
* the need for surgical treatment during follow-up,
* the deterioration of tear anatomy (tear size, muscle atrophy, fatty degeneration) during follow-up
* the actual clinical shoulder condition (as given by shoulder scores) at reexamination.

Study purpose: We want to assess the anatomic and clinical long-term results of physiotherapy for potentially repairable rotator cuff tears. We want to find out if tear anatomy of unrepaired rotator cuff tears deteriorates over time and if such a deterioration is associated with a development of more serious degrees of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Full-thickness rotator cuff tear diagnosed between 2002 and 2005 by both sonography and MRI.

At the time of diagnosis (2002 to 2005):

* Typical clinical symptoms for a rotator cuff tear including pain laterally on upper humerus, painful arc, positive impingement test (Neer or Hawkins)
* Potentially repairable tear (tear size up to 3 cm, muscle atrophy not exceeding grade 2 according to Thomazeau, fatty degeneration not exceeding grade 1 according to Goutallier).
* Treated by physiotherapy for at least 3 months

Exclusion Criteria:

At the time of diagnosis (2002 to 2005):

* Full-thickness tears of the subscapularis tendon or of the entire supraspinatus and infraspinatus tendons
* Other symptomatic shoulder pathology including long head of the biceps tendon pathology, acromioclavicular joint pathology, shoulder instability, inflammatory diseases, glenohumeral arthritis
* Earlier treated with rotator cuff repair in the study shoulder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with a symptomatic full-thickness rotator cuff tear in the period 2002 to 2005. All tears were deemed to be repairable at the time of the diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2012-03; Primary Completion 2016-02 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Shoulder sonography | Baseline to 8-10 years follow-up
  Sonographic shoulder examination was performed for all study patients before treatment was given. All patients will be reexamined by sonography after 8 to 10 years. The finding of interest is the change of tear size as determined by sonography

SECONDARY OUTCOMES:
Number of relapses during follow-up | 8 to 10 years
  At follow-up patients have to report how many new periods with shoulder pain they have experienced since the time of diagnosis
Number of patients who needed surgical treatment of their shoulder during follow-up | 8 to 10 years
  At follow-up, patients have to report the number of surgical interventions in their study shoulder since the time of diagnosis.
MRI of the shoulder | MRI will be performed at 8 to 10 years follow-up
  At the time of diagnosis, no patient had serious muscle atrophy or fatty degeneration as determined by MRI. The finding of interest at 8 to 10 years follow-up is the number of patients who have progressed to serious muscle atrophy or fatty degeneration during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Moosmayer, MD, PhD, Principal Investigator — Vestre Viken Hospital Trust
Locations (1):
- Martina Hansen's Hospital, Sandvika, Norway

REFERENCES:
- [Result] Moosmayer S, Gartner AV, Tariq R. The natural course of nonoperatively treated rotator cuff tears: an 8.8-year follow-up of tear anatomy and clinical outcome in 49 patients. J Shoulder Elbow Surg. 2017 Apr;26(4):627-634. doi: 10.1016/j.jse.2016.10.002. Epub 2017 Jan 12. PMID 28089257